CLINICAL TRIAL: NCT02412046
Title: Quantification of the Pressure Threshold Related to Tissue Injury in Bedriden Paraplegics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the PhD in charge of the study
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 95022
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Pressure Ulcer; Bedsore; Spinal Cord Injury; Paraplegia
Keywords: Pressure ulcer; Interface pressure; Pressure mapping device; Ischemia reperfusion; Monitoring; Microvascularization
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Time of the first biopsy: H0 (Active Comparator): For the patients in arm H0, the first biopsy is done as soon as the patient is lying on the air mattress.
  Interventions: Procedure: Muscle biopsy
- Time of the first biopsy: H1 (Active Comparator): For a patient in arm H1, it is done after 1 hour lying on the air mattress.
  Interventions: Procedure: Muscle biopsy
- Time of the first biopsy: H2 (Active Comparator): For a patient in arm H2, it is done after 2 hour lying on the air mattress.
  Interventions: Procedure: Muscle biopsy
- Time of the first biopsy: H3 (Active Comparator): For a patient in arm H3, it is done after 3 hour lying on the air mattress.
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy

SUMMARY:
The aim of this study is to correlate the intensity and the duration of a mechanical strain, applied over the skin of a bedridden paraplegics, with the microvascularization parameters (oxygen saturation, blood flow and blood volume) and the early inflammatory mechanism. We want to detect the early stage of irreversible damage for each patient. To achieve this goal, we measure some specifics data over a group of 48 paraplegics admitted in the hospital for a pressure ulcer surgical treatment. The patients are randomly distributed in 4 groups. First the interface pressure between the patient body and the air mattress is recorded continuously for 3 hours (= the repositioning patient frequency): we have the pressure over each point of the patient body in contact with the mattress on this time lap. Then, we will measure the microvascularization parameters, using an O2C medical device over a trochanter on a specific anatomical area which will be thereafter biopsied. Finally, depending on the group in which they were randomly distributed, the patient will undergo a muscle biopsy on his or her trochanter at 0h, 1h, 2h or 3h after they lie down on the air mattress. This way, we will be able to determine the effect of the mechanical strain duration on the physiologic parameters. The following day, the patient is undergoing his or her surgery for removing the necrotic area of the bedsore. At the same time, we will recover some of the sample near the bedsore which would serve as a maximum inflammatory response. Then a second muscle biopsy will be performed on an innervated area to be able to determine a basal concentration of biomarkers.

The inclusion period for this study will be 3 years. All the patients are followed for 24 hours then they will be followed by medical staff in their bedsore resection setting.

The data gained for this study will hopefully help the scientific world to achieve a better understanding of the pressure ulcer aetiology. They will also be helpful to achieve a mobilization of the patient specific of his or her inherent characteristics with a high sensitivity level. This way we will have a more efficient bedsore prevention.

ELIGIBILITY:
Inclusion Criteria:

* Educated consent signed,
* Older than 18,
* Paraplegia for at least 6 months,
* Patient's Body Mass Index > 18,5kg/m²,
* Surgery planned for pressure ulcer resection,
* Pressure Ulcer classification (EPUAP) at least III or IV

Exclusion Criteria:

* Cardiac pathology,
* Duchenne muscular dystrophy,
* Dementia,
* Presence of a tumourous wound,
* Stade IV arteritis non-revascularisable,
* Diabetes mellitus,
* Cachexia,
* Impossibility to stop the anti-coagulant treatment 24 hours before the patient admission,
* Xylocaine allergy,
* Patient took aspirin or anti-inflammatory 3 days before the biopsy,
* Patient taking part in another study,
* Patient with no health insurance,
* Pregnant women or breast-feeding, patient unable to give his or her educated consent, ward of the state (art. L.1121-6, L.1121-7, L.1211-8, L.1211-9)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
The interface pressure will be continuously assessed using a mapping device (XSensor) during 3 hours. | The first day of the patient admission (during the first 3 hours).

SECONDARY OUTCOMES:
The microvascularization changes underneath the compressed skin and the inflammatory response of the muscle cells. | The first day of the patient admission (during the first 3 hours).
  The blood flow, the oxygen saturation and the hemoglobin amount will be measured using a medical device called Oxygen To See (O2C). The reactive oxygen species or ROS and other specific biomarkers will be used to measure and quantify the inflammatory response of muscle cells.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France